CLINICAL TRIAL: NCT03541538
Title: Hypoalgesic Effects of Specific vs Non-specific Cervical Manipulation in Healthy Subjects
Brief Title: Hypoalgesic Effect of Cervical Manipulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Jonathan Daniel Telles, Principal Investigator, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: U1111-1214-1243
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Pain
Keywords: joint manipulation; cervical; pressure pain; manual therapy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Participants received two interventions randomly at two times: global manipulation (GM) and specific manipulation (MS)
Who Masked: Participant, Outcomes Assessor
Masking Description: Examiner 1 will receive the blinding outcome will be asked: "Which intervention does the patienth as received: global manipulation or especific manipulation" Their responses to these questions will be recorded and used to measure the adequacy of participants and examiners.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Global manipulation (Active Comparator): Manual therapy performed in the cervical region in a non-specific way.
  Interventions: Device: Global manipulation
- Especific manipulation (Experimental): manual therapy performed specifically on the C6-7 segment
  Interventions: Device: Especific manipulation

INTERVENTIONS:
Device: Global manipulation — The therapist positioned himself at the head of the stretcher and with one hand supported the side of the participant's face. With the other hand supported the opposite face of the same and then performed contralateral rotation of the cervical and a slight traction to the tissue barrier to perform the manipulation impulse of high speed and short amplitude in rotation. The procedure was carried out bilaterally.
  Arms: Global manipulation
Device: Especific manipulation — The therapist positioned himself at the head of the stretcher and with one hand kept the middle phalange of the second finger laterally on the articular processes of the C6-7 vertebrae. With the contralateral hand he supported the opposing face of the participant by performing a tilt up to the C6-7 segment and contralateral rotation up to the tissue barrier to carry out the impulse quickly and short. The procedure was carried out bilaterally.
  Arms: Especific manipulation

SUMMARY:
This study evaluates the hypoalgesic effect of global and specific cervical joint manipulation in healthy individuals. At first the participants received one of the interventions and after 48 hours, the other.

DETAILED DESCRIPTION:
Cervical Joint Manipulation (CJM) are often used for pain treatment.

Joint manipulation generates a series of stimuli within the central nervous system through the activation of proprioceptors located in the joint capsule or muscles, stimulates the PAG, causing pain inhibition by activation of non-opioid descending inhibitory pathways.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects of both sexes
* without pain complaints in the last 90 days

Exclusion Criteria:

* previous spinal surgeries
* spinal canal stenosis
* vertebral fracture
* spondylolisthesis
* cancer
* acute infections
* hemorrhagic disorders
* active tuberculosis
* deep vein thrombosis
* osteoporosis
* rheumatic diseases
* metabolic diseases
* cardiorespiratory diseases
* smoking injury
* musculoskeletal injury
* use of pacemaker
* women in menstrual period
* pregnant women
* use of pain-killers in the last 48 hours
* use of anti-inflammatory drugs in the last 48 hours
* previous joint manipulation treatments
* aversion to cervical joint manipulation
* positivity in the vertebral artery test
* headache in the last seven days

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold at the posterior region of the forearm | 1 minute after the end of the intervention.
  The subjects were placed supine on a stretcher with their elbows fully extended and the anterior portion of the forearm resting on the stretcher. Subjects were instructed to keep their eyes closed during attempts. The examiner used a Somedic Type II digital pressure algometer (Somedic Inc, Hörby, Sweden) on the posterior region of the forearm 10cm below the lateral epicondyle of the elbow towards the third finger, keeping the forearm in pronation. The pressure was then applied perpendicular to the skin at a rate of 40kPa / s using a 1cm2 flat circular probe covered with 1mm of rubber to prevent any skin pain caused by sharp metal edges.

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Liebano, Dr., Principal Investigator — Universidade Federal de São Carlos - UFScar
Locations (1):
- Ufscar - Universidade Federal de São Carlos, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Achalandabaso A, Plaza-Manzano G, Lomas-Vega R, Martinez-Amat A, Camacho MV, Gasso M, Hita-Contreras F, Molina F. Tissue damage markers after a spinal manipulation in healthy subjects: a preliminary report of a randomized controlled trial. Dis Markers. 2014;2014:815379. doi: 10.1155/2014/815379. Epub 2014 Dec 25. PMID 25609853
- [Background] Almay BG, Johansson F, von Knorring L, Sakurada T, Terenius L. Long-term high frequency transcutaneous electrical nerve stimulation (hi-TNS) in chronic pain. Clinical response and effects on CSF-endorphins, monoamine metabolites, substance P-like immunoreactivity (SPLI) and pain measures. J Psychosom Res. 1985;29(3):247-57. doi: 10.1016/0022-3999(85)90051-0. PMID 2411923
- [Background] Bergmann TF. Short lever, specific contact articular chiropractic technique. J Manipulative Physiol Ther. 1992 Nov-Dec;15(9):591-5. PMID 1469343
- [Background] Bialosky JE, Bishop MD, Price DD, Robinson ME, George SZ. The mechanisms of manual therapy in the treatment of musculoskeletal pain: a comprehensive model. Man Ther. 2009 Oct;14(5):531-8. doi: 10.1016/j.math.2008.09.001. Epub 2008 Nov 21. PMID 19027342
- [Background] Bicalho E, Setti JA, Macagnan J, Cano JL, Manffra EF. Immediate effects of a high-velocity spine manipulation in paraspinal muscles activity of nonspecific chronic low-back pain subjects. Man Ther. 2010 Oct;15(5):469-75. doi: 10.1016/j.math.2010.03.012. Epub 2010 May 5. PMID 20447857
- [Background] Bishop MD, Beneciuk JM, George SZ. Immediate reduction in temporal sensory summation after thoracic spinal manipulation. Spine J. 2011 May;11(5):440-6. doi: 10.1016/j.spinee.2011.03.001. Epub 2011 Apr 3. PMID 21463970
- [Background] Boal RW, Gillette RG. Central neuronal plasticity, low back pain and spinal manipulative therapy. J Manipulative Physiol Ther. 2004 Jun;27(5):314-26. doi: 10.1016/j.jmpt.2004.04.005. PMID 15195039
- [Background] Coronado RA, Gay CW, Bialosky JE, Carnaby GD, Bishop MD, George SZ. Changes in pain sensitivity following spinal manipulation: a systematic review and meta-analysis. J Electromyogr Kinesiol. 2012 Oct;22(5):752-67. doi: 10.1016/j.jelekin.2011.12.013. Epub 2012 Jan 30. PMID 22296867
- [Background] Costa LO, Maher CG, Latimer J, Ferreira PH, Ferreira ML, Pozzi GC, Freitas LM. Clinimetric testing of three self-report outcome measures for low back pain patients in Brazil: which one is the best? Spine (Phila Pa 1976). 2008 Oct 15;33(22):2459-63. doi: 10.1097/BRS.0b013e3181849dbe. PMID 18923324
- [Background] Dailey DL, Rakel BA, Vance CGT, Liebano RE, Amrit AS, Bush HM, Lee KS, Lee JE, Sluka KA. Transcutaneous electrical nerve stimulation reduces pain, fatigue and hyperalgesia while restoring central inhibition in primary fibromyalgia. Pain. 2013 Nov;154(11):2554-2562. doi: 10.1016/j.pain.2013.07.043. Epub 2013 Jul 27. PMID 23900134
- [Background] Descarreaux M, Blouin JS, Drolet M, Papadimitriou S, Teasdale N. Efficacy of preventive spinal manipulation for chronic low-back pain and related disabilities: a preliminary study. J Manipulative Physiol Ther. 2004 Oct;27(8):509-14. doi: 10.1016/j.jmpt.2004.08.003. PMID 15510094
- [Background] Degenhardt BF, Darmani NA, Johnson JC, Towns LC, Rhodes DC, Trinh C, McClanahan B, DiMarzo V. Role of osteopathic manipulative treatment in altering pain biomarkers: a pilot study. J Am Osteopath Assoc. 2007 Sep;107(9):387-400. PMID 17908831
- [Background] Dishman JD, Cunningham BM, Burke J. Comparison of tibial nerve H-reflex excitability after cervical and lumbar spine manipulation. J Manipulative Physiol Ther. 2002 Jun;25(5):318-25. doi: 10.1067/mmt.2002.124420. PMID 12072852
- [Background] DeVocht JW, Pickar JG, Wilder DG. Spinal manipulation alters electromyographic activity of paraspinal muscles: a descriptive study. J Manipulative Physiol Ther. 2005 Sep;28(7):465-71. doi: 10.1016/j.jmpt.2005.07.002. PMID 16182019
- [Background] Dunning J, Rushton A. The effects of cervical high-velocity low-amplitude thrust manipulation on resting electromyographic activity of the biceps brachii muscle. Man Ther. 2009 Oct;14(5):508-13. doi: 10.1016/j.math.2008.09.003. Epub 2008 Nov 21. PMID 19027344
- [Background] Fernandez-de-Las-Penas C. Clinical evaluation of cervicogenic headache: a clinical perspective. J Man Manip Ther. 2008;16(2):81. doi: 10.1179/106698108790818440. No abstract available. PMID 19119391
- [Background] Fernandez-de-Las-Penas C, Alonso-Blanco C, Cleland JA, Rodriguez-Blanco C, Alburquerque-Sendin F. Changes in pressure pain thresholds over C5-C6 zygapophyseal joint after a cervicothoracic junction manipulation in healthy subjects. J Manipulative Physiol Ther. 2008 Jun;31(5):332-7. doi: 10.1016/j.jmpt.2008.04.006. PMID 18558274
- [Background] Fernandez-de-las-Penas C, Perez-de-Heredia M, Brea-Rivero M, Miangolarra-Page JC. Immediate effects on pressure pain threshold following a single cervical spine manipulation in healthy subjects. J Orthop Sports Phys Ther. 2007 Jun;37(6):325-9. doi: 10.2519/jospt.2007.2542. PMID 17612359
- [Background] Flynn TW, Childs JD, Fritz JM. The audible pop from high-velocity thrust manipulation and outcome in individuals with low back pain. J Manipulative Physiol Ther. 2006 Jan;29(1):40-5. doi: 10.1016/j.jmpt.2005.11.005. PMID 16396728
- [Background] Gay CW, Robinson ME, George SZ, Perlstein WM, Bishop MD. Immediate changes after manual therapy in resting-state functional connectivity as measured by functional magnetic resonance imaging in participants with induced low back pain. J Manipulative Physiol Ther. 2014 Nov-Dec;37(9):614-27. doi: 10.1016/j.jmpt.2014.09.001. Epub 2014 Oct 3. PMID 25284739
- [Background] George SZ, Bishop MD, Bialosky JE, Zeppieri G Jr, Robinson ME. Immediate effects of spinal manipulation on thermal pain sensitivity: an experimental study. BMC Musculoskelet Disord. 2006 Aug 15;7:68. doi: 10.1186/1471-2474-7-68. PMID 16911795
- [Background] Jordon MK, Beattie PF, D'Urso S, Scriven S. Spinal manipulation does not affect pressure pain thresholds in the absence of neuromodulators: a randomized controlled trial. J Man Manip Ther. 2017 Sep;25(4):172-181. doi: 10.1080/10669817.2016.1230352. Epub 2016 Sep 12. PMID 28912629
- [Background] Korr IM. Proprioceptors and somatic dysfunction. J Am Osteopath Assoc. 1975 Mar;74(7):638-50. No abstract available. PMID 124754
- [Background] Leffler AS, Hansson P, Kosek E. Somatosensory perception in a remote pain-free area and function of diffuse noxious inhibitory controls (DNIC) in patients suffering from long-term trapezius myalgia. Eur J Pain. 2002;6(2):149-59. doi: 10.1053/eujp.2001.0312. PMID 11900475
- [Background] Leffler AS, Hansson P, Kosek E. Somatosensory perception in patients suffering from long-term trapezius myalgia at the site overlying the most painful part of the muscle and in an area of pain referral. Eur J Pain. 2003;7(3):267-76. doi: 10.1016/S1090-3801(02)00138-6. PMID 12725850
- [Background] Liebano RE, Rakel B, Vance CGT, Walsh DM, Sluka KA. An investigation of the development of analgesic tolerance to TENS in humans. Pain. 2011 Feb;152(2):335-342. doi: 10.1016/j.pain.2010.10.040. Epub 2010 Dec 8. PMID 21144659
- [Background] Liebano RE, Vance CG, Rakel BA, Lee JE, Cooper NA, Marchand S, Walsh DM, Sluka KA. Transcutaneous electrical nerve stimulation and conditioned pain modulation influence the perception of pain in humans. Eur J Pain. 2013 Nov;17(10):1539-46. doi: 10.1002/j.1532-2149.2013.00328.x. Epub 2013 May 6. PMID 23650092
- [Background] Malisza KL, Gregorash L, Turner A, Foniok T, Stroman PW, Allman AA, Summers R, Wright A. Functional MRI involving painful stimulation of the ankle and the effect of physiotherapy joint mobilization. Magn Reson Imaging. 2003 Jun;21(5):489-96. doi: 10.1016/s0730-725x(03)00074-2. PMID 12878258
- [Background] Nakatsuka T, Chen M, Takeda D, King C, Ling J, Xing H, Ataka T, Vierck C, Yezierski R, Gu JG. Substance P-driven feed-forward inhibitory activity in the mammalian spinal cord. Mol Pain. 2005 Jun 29;1:20. doi: 10.1186/1744-8069-1-20. PMID 15987503
- [Background] Nussbaum EL, Downes L. Reliability of clinical pressure-pain algometric measurements obtained on consecutive days. Phys Ther. 1998 Feb;78(2):160-9. doi: 10.1093/ptj/78.2.160. PMID 9474108
- [Background] de Oliveira RF, Liebano RE, Costa Lda C, Rissato LL, Costa LO. Immediate effects of region-specific and non-region-specific spinal manipulative therapy in patients with chronic low back pain: a randomized controlled trial. Phys Ther. 2013 Jun;93(6):748-56. doi: 10.2522/ptj.20120256. Epub 2013 Feb 21. PMID 23431209
- [Background] Molina-Ortega F, Lomas-Vega R, Hita-Contreras F, Plaza Manzano G, Achalandabaso A, Ramos-Morcillo AJ, Martinez-Amat A. Immediate effects of spinal manipulation on nitric oxide, substance P and pain perception. Man Ther. 2014 Oct;19(5):411-7. doi: 10.1016/j.math.2014.02.007. Epub 2014 Mar 5. PMID 24674816
- [Background] Pickar JG. Neurophysiological effects of spinal manipulation. Spine J. 2002 Sep-Oct;2(5):357-71. doi: 10.1016/s1529-9430(02)00400-x. PMID 14589467
- [Background] Pickar JG, Wheeler JD. Response of muscle proprioceptors to spinal manipulative-like loads in the anesthetized cat. J Manipulative Physiol Ther. 2001 Jan;24(1):2-11. doi: 10.1067/mmt.2001.112017. PMID 11174689
- [Background] Schneider M. Changes in pressure pain sensitivity in latent myofascial trigger points in the upper trapezius muscle after a cervical spine manipulation in pain-free subjects. J Manipulative Physiol Ther. 2008 Mar;31(3):251; author reply 251-2. doi: 10.1016/j.jmpt.2008.02.011. No abstract available. PMID 18394505
- [Background] Savva C, Giakas G, Efstathiou M. The role of the descending inhibitory pain mechanism in musculoskeletal pain following high-velocity, low amplitude thrust manipulation: a review of the literature. J Back Musculoskelet Rehabil. 2014;27(4):377-82. doi: 10.3233/BMR-140472. PMID 24867897
- [Background] Sluka KA, Deacon M, Stibal A, Strissel S, Terpstra A. Spinal blockade of opioid receptors prevents the analgesia produced by TENS in arthritic rats. J Pharmacol Exp Ther. 1999 May;289(2):840-6. PMID 10215661
- [Background] Sluka KA, Wright A. Knee joint mobilization reduces secondary mechanical hyperalgesia induced by capsaicin injection into the ankle joint. Eur J Pain. 2001;5(1):81-7. doi: 10.1053/eujp.2000.0223. PMID 11394925
- [Background] Staud R. Treatment of fibromyalgia and its symptoms. Expert Opin Pharmacother. 2007 Aug;8(11):1629-42. doi: 10.1517/14656566.8.11.1629. PMID 17685881
- [Background] Treede RD, Rief W, Barke A, Aziz Q, Bennett MI, Benoliel R, Cohen M, Evers S, Finnerup NB, First MB, Giamberardino MA, Kaasa S, Kosek E, Lavand'homme P, Nicholas M, Perrot S, Scholz J, Schug S, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ. A classification of chronic pain for ICD-11. Pain. 2015 Jun;156(6):1003-1007. doi: 10.1097/j.pain.0000000000000160. No abstract available. PMID 25844555
- [Background] Vicenzino B, Collins D, Benson H, Wright A. An investigation of the interrelationship between manipulative therapy-induced hypoalgesia and sympathoexcitation. J Manipulative Physiol Ther. 1998 Sep;21(7):448-53. PMID 9777544
- [Background] Vigotsky AD, Bruhns RP. Corrigendum to "The Role of Descending Modulation in Manual Therapy and Its Analgesic Implications: A Narrative Review". Pain Res Treat. 2017;2017:1535473. doi: 10.1155/2017/1535473. Epub 2017 Oct 26. PMID 29225969
- [Background] Walton DM, Macdermid JC, Nielson W, Teasell RW, Chiasson M, Brown L. Reliability, standard error, and minimum detectable change of clinical pressure pain threshold testing in people with and without acute neck pain. J Orthop Sports Phys Ther. 2011 Sep;41(9):644-50. doi: 10.2519/jospt.2011.3666. Epub 2011 Sep 1. PMID 21885906
- [Background] Wassinger CA, Rich D, Cameron N, Clark S, Davenport S, Lingelbach M, Smith A, Baxter GD, Davidson J. Cervical & thoracic manipulations: Acute effects upon pain pressure threshold and self-reported pain in experimentally induced shoulder pain. Man Ther. 2016 Feb;21:227-32. doi: 10.1016/j.math.2015.08.009. Epub 2015 Aug 28. PMID 26391291
- [Background] Welch A, Boone R. Sympathetic and parasympathetic responses to specific diversified adjustments to chiropractic vertebral subluxations of the cervical and thoracic spine. J Chiropr Med. 2008 Sep;7(3):86-93. doi: 10.1016/j.jcm.2008.04.001. PMID 19646369
- [Background] Wright A. Hypoalgesia post-manipulative therapy: a review of a potential neurophysiological mechanism. Man Ther. 1995 Nov;1(1):11-6. doi: 10.1054/math.1995.0244. PMID 11327789
- See also: La Société Française de Médecine Manuelle — https://www.sofmmoo.org/documents/mode_action_mv_jym-pv.pdf